CLINICAL TRIAL: NCT05043558
Title: The Protective Effect of Prostaglandin on Coronary Microcirculation and Ventricular Remodeling After Reperfusion Therapy in Acute ST-segment Elevation Myocardial Infarction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LHD Beraprost sodium
Record Dates: First submitted 2021-08-25; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: STEMI
Keywords: Beprostaglandin sodium
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beprostaglandin sodium (Experimental)
  Interventions: Drug: beprostaglandin sodium
- control group (No Intervention)

INTERVENTIONS:
Drug: beprostaglandin sodium — beprostaglandin sodium
  Arms: beprostaglandin sodium

SUMMARY:
To explore the protective effect of prostaglandin sodium on coronary microcirculation function and ventricular remodeling after reperfusion treatment of acute ST-segment elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* 1) Meet the diagnostic criteria for acute ST-segment elevation myocardial infarction: ①The onset of ischemic chest pain lasts for more than 30 minutes and cannot be relieved by taking nitroglycerin; ②The ECG has two or more ST-segment elevations in adjacent leads , Limb leads ≥ 1mm, pectoral leads ≥ 2mm; or newly-appearing left bundle branch block; ③The increase in serum markers of myocardial necrosis is at least twice the normal value; (2) Coronary angiography confirmed acute myocardial infarction; (3) Direct PCI treatment within 12 hours of onset; (4) Complete clinical and radiographic data.

Exclusion Criteria:

* (1) Those who do not cooperate in the inspection, have poor compliance, and cannot guarantee the completion of the test; (2) Persons with consciousness impairment, obvious intellectual impairment and mental abnormality; (3) With metal foreign bodies, such as metal prostheses, intraocular metal foreign bodies, intracranial aneurysm clamps, etc.; (4) Those who suffer from closure phobia; (5) Those who have had a history of myocardial infarction, PCI treatment, or coronary artery bypass graft; (6) Factors affecting the changes in the ST segment of the electrocardiogram: complete left bundle branch block, pre-excitation syndrome, pacemaker electrocardiogram

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-01-10 (Estimated); Study Completion 2022-01-12 (Estimated)

PRIMARY OUTCOMES:
ultrasound and CMR to assess the characteristics of myocardial infarction | 3 years
  Q-LAB Scale Scale calculation score

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People' S Hospital, Shenzhen, Guangdong, China